CLINICAL TRIAL: NCT05581979
Title: PSMA-PET Imaging of Salivary Gland Tumours and Other Rare Cancers
Status: Completed | Type: Observational
Sponsor: National Cancer Centre, Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: PSMA 01
Record Dates: First submitted 2022-09-28; First posted 2022-10-17 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Salivary Gland Tumor; Rare Malignant Neoplasm
Keywords: 68-Ga PSMA PET Imaging; Salivary Gland; Radiolabeling; Gallium-68; PET scan; Prostate Specific Membrane Antigen; Adenocystic Carcinoma; Rare Tumours
MeSH Terms: conditions — Salivary Gland Neoplasms; Carcinoma, Adenoid Cystic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 68-Ga PSMA PET scan: 68-Ga PSMA PET scan
  Interventions: Diagnostic Test: 68-Ga PSMA PET scan

INTERVENTIONS:
Diagnostic Test: 68-Ga PSMA PET scan — On the scheduled visit date for the study,
  * An intravenous cannula (plug) will be inserted in a vein in the participant's arm, through which the 68-Ga PSMA radiotracer for the scan will be injected. The infusion will take about 1-2 minutes.
  * PET imaging will be performed with a dedicated PET/CT scanner. 2.5-6.0 mCi (depending on weight of the patient) of PSMA radiotracer will be injected intravenously.

SUMMARY:
The objectives of this pilot feasibility study, which is on the use of 68-Ga PSMA PET imaging of salivary gland tumours, are

* to determine the proportion of patients with high PSMA-ligand uptake on Ga-68 PSMA imaging in locally advanced, recurrent or metastatic salivary gland cancers and other rare cancer; and
* to determine if in vitro PSMA expression correlates to PSMA-ligand uptake on Ga-68 PSMA imaging in locally advanced, recurrent or metastatic salivary gland cancers and other rare cancers.

The hypotheses of this study are that there is high PSMA-ligand uptake on Ga-68 PSMA imaging in locally advanced, recurrent or metastatic salivary gland cancers and other rare cancers; and that in vitro PSMA expression correlates to PSMA-ligand uptake on Ga-68 PSMA imaging.

DETAILED DESCRIPTION:
The potential participant will be screened and confirmed for eligibility by the appropriate study-team member. A signed IRB approved informed consent will be obtained prior to conducting any study-related procedures.

On the scheduled visit date for the study,

* An intravenous cannula (plug) will be inserted in a vein in the participant's arm, through which the 68-Ga PSMA radiotracer for the scan will be injected. The infusion will take about 1-2 minutes.
* PET imaging will be performed with a dedicated PET/CT scanner. 2.5-6.0 mCi (depending on weight of the patient) of PSMA radiotracer will be injected intravenously.
* A PET scan will be done around 60 minutes after the injection of the 68-Ga PSMA imaging agent.
* During imaging, the participant will be asked to lie still and may be asked to hold his/her breath for a few seconds.
* Imaging will be performed using a PET/CT, which will take 30 to 40 minutes to complete. Imaging of the body from vertex to mid thigh or feet will be obtained.
* After the completion of the scan, the plug will be removed.

A Final Study Visit will take place on that one scheduled day. The participant will not need to visit the doctor's office during the course of the study outside of their usual scheduled doctor's follow up appointments.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced, metastatic or locally recurrent salivary gland cancers OR rare cancers (Examples of rare cancers: thyroid ca, cholangio ca, pancreatic ca, gall bladder ca, sarcoma)
* Sample of biopsied tissue available for analysis
* Histologically confirmed diagnoses
* Above 21 years of age
* Able to provide informed consent

Exclusion Criteria:

* Those who do not meet above inclusion criteria
* Diagnosis of haematological malignancies
* Patients with more than one cancer diagnosis
* Contraindication to 68Ga-PSMA PET/CT

  * E.g.: pregnant patients, breast feeding patients, renal impairment, liver impairment, allergy to components of the test
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow up schedule
* Ongoing participation in any other clinical trial

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients would have to have histologically confirmed diagnoses, are above 21 years of age, have no contraindication to 68Ga-PSMA PET/CT and able to give consent.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2022-01-26 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
The proportion of patients with high PSMA-ligand uptake on Ga-68 PSMA imaging in locally advanced, recurrent or metastatic salivary gland cancers and other rare cancer. | Through study completion, to June 2024.
  The proportion of patients with PSMA-ligand uptake greater than liver uptake on Ga-68 PSMA imaging in locally advanced, recurrent or metastatic salivary gland cancers and other rare cancer.

SECONDARY OUTCOMES:
Correlation between in vitro PSMA expression and PSMA-ligand uptake on Ga-68 PSMA imaging in locally advanced, recurrent or metastatic salivary gland cancers and other rare cancers. | Through study completion, to June 2024.
  Correlation between the value of IHC PSMA expression and the PSMA PET SUVmax in locally advanced, recurrent or metastatic salivary gland cancers and other rare cancers.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Wen-Long NEI, MD, Principal Investigator — National Cancer Centre, Singapore
Locations (1):
- National Cancer Centre Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided